CLINICAL TRIAL: NCT03387891
Title: Clinical Testing on Newly Developed Monitoring Technology (The Cortrium C3 Device) for Continuous Measurements of ECG, Respiratory Rate, Body Surface Temperature and Accelerometer Data for Patients With Cancer
Brief Title: Clinical Testing of the Cortrium C3 Device
Status: Completed | Type: Observational
Sponsor: Cortrium (Industry)
Collaborators: University College Absalon (Other)
Responsible Party: Sponsor
Other Study IDs: 94.1.05-5660-10728
Record Dates: First submitted 2017-04-30; First posted 2018-01-02 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients: Cancer patients admitted to hospital for treatment or monitoring of health condition
  Interventions: Device: Cortrium C3 device

INTERVENTIONS:
Device: Cortrium C3 device — Paired measurements of data from C3 device with golden standard methods or equipment

SUMMARY:
Clinical data validation of the C3 device as a Vital Sign Monitoring System for patients under cancer treatment.

DETAILED DESCRIPTION:
Cortrium has developed the C3 device. The C3 device contains sensors that monitors Electrocardiogram (ECG), Respiratory rate (breathes per minute), and Body surface temperature. Also, the C3 device contains an accelerometer for registration of the body posture.

The following thesis will be tested:

Thesis 1) Pulse: The C3 device produces clinically validated pulse data. Thesis 2) Respiratory rate: The C3 device produces clinically validated respiratory rate data (breaths per minute). Thesis 3) Infection: With no justified statistical significant correlation between skin and body temperature, the study is exploring how to prevent aggravated or lethal outcomes of cancer treatment, e.g. chemotherapy, by using vital signs measurements combined with accelerometer data to detect infection levels. Thesis 4) The qualitative study: The study will report the advantages and disadvantages regarding new technological solutions, and the change in workflow and healthcare provision as it is experienced by the healthcare personnel and the patients. The data validation studies (thesis 1-3) will be tested in comparison with golden standard measurements methods and/or data validated medical equipment.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent persons - i.e., patients considered able to understand the information given about the clinical trial
* Person is 18 years or older
* Person has given a written informed consent

Exclusion Criteria:

* Not legally competent patients
* Pregnant and lactating women
* Fertile women, who do not use contraceptives
* Patients under 18 years
* Patients with known heart-related disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer diagnose admitted to the hospital for treatment and/or monitoring of their health condition.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Pulse rate | May 2017-March 2018
  Continuous measurements from C3 device. Punctual measurement observed by the healthcare personnel
Respiratory rate | May 2017-March 2018
  Continuous measurements from C3 device. Punctual measurement observed by the

SECONDARY OUTCOMES:
Infection | May 2017-March 2018
  Exploratory study - Comparison of all sensors embedded within the C3 device to the patient infection level (measured as fever)
Design & Workflow studies | May 2017-March 2018
  Observational studies and interviews with healthcare personnel and patients regarding the C3 device.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Eric Nielsen, COO, Study Chair — Cortrium
Locations (1):
- University Medical Center Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data will be available for workflow design and nurse studies.